CLINICAL TRIAL: NCT03068208
Title: Efficacy of Methylene Blue Mediated Photodynamic Therapy for Primary Localized Cutaneous Amyloidosis Treatment in Asians: Pilot Study
Brief Title: Efficacy of Methylene Blue Mediated Photodynamic Therapy for Primary Localized Cutaneous Amyloidosis Treatment in Asians
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Chulalongkorn University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CU_MBPDT_for_amyloidosis
Record Dates: First submitted 2017-02-20; First posted 2017-03-01 (Actual); Last update posted 2017-03-01 (Actual); Status verified 2017-02

CONDITIONS: Lichen Amyloidosis
Keywords: Methylene blue; photodynamic therapy; primary cutaneous localized amyloidosis; lichen amyloidosis
MeSH Terms: conditions — Amyloidosis, Primary Cutaneous

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MB-PDT (Experimental)
  Interventions: Procedure: Methylene blue-mediated photodynamic therapy
- Control (No Intervention)

INTERVENTIONS:
Procedure: Methylene blue-mediated photodynamic therapy — The 2% MB aqueous solution was applied to the lesion until saturation occurred, followed by a occlusive dressing and rest period of 30 minutes. After the rest period, the lesion was immediately illuminated with incoherent red light (peak emission spectrum at 630-640 nm)
  Arms: MB-PDT

SUMMARY:
Efficacy of Methylene blue mediated Photodynamic therapy for primary localized cutaneous amyloidosis treatment in Asians, pilot study.

ELIGIBILITY:
Inclusion Criteria:

* Patients, aged > 18 years old with lichen amyloidosis diagnosed by using clinical presentation and pathological findings.

Exclusion Criteria:

* Those with systemic disease associated cutaneous amyloidosis
* Pregnancy or lactating woman
* Those who are allergic to urea, olive oil
* Those who are photosensitive to ultraviolet radiation
* Those who had been previously treated with any of which -medications, radiation, laser within 3 months and 1 month for topical therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2017-05-01 (Estimated); Primary Completion 2018-04-30 (Estimated); Study Completion 2018-06-30 (Estimated)

PRIMARY OUTCOMES:
Roughness evaluation by using visioscan | Change from baseline roughness at every 2 weeks up to 16 weeks
  The improvement of roughness during the treatment

CONTACTS AND LOCATIONS:
Overall Officials: Einapak Amnarttrakul, M.D., Principal Investigator — Chulalongkorn University
Locations (1):
- King Chulalongkorn Memorial Hospital, Bangkok, Bangkok, Thailand

IPD SHARING:
Plan to Share IPD: Undecided